CLINICAL TRIAL: NCT05352217
Title: The Possible Influence of Different Follow-up Modalities on Overall Survival in Ovarian Cancer: A Multicenter Observational Cohort Study
Brief Title: The Possible Influence of Different Follow-up Modalities on Overall Survival in Ovarian Cancer
Acronym: ECOvar
Status: Terminated | Type: Observational
Why Stopped: Accrual rate fell far below needed accrual rate.
Sponsor: Stiftung Swiss Tumor Institute (Other)
Collaborators: Klinik Hirslanden, Zurich (Other); Manja Gideon Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-D0052
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Patient Reported Outcome Measures; Ovarian Neoplasms
Keywords: ePRO; PRO; Electronic Patient Reported Outcome; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mobile app ovarian cancer followup (ePRO) — The study is designed as an observational cohort study, aiming to evaluate, whether a structured recording of symptoms by a mobile app contributes insight in the follow-up modalities of ovarian cancer patients.

SUMMARY:
The study is designed as an observational cohort study, aiming to evaluate, whether a structured recording of symptoms by a mobile app contributes insight in the follow-up modalities of ovarian cancer patients.

DETAILED DESCRIPTION:
The observational study will examine different follow-up modalities for ovarian cancer patients with the ultimate goal of improving follow-up strategies for an improved well-being and better clinical outcomes. The primary objective is to quantify the effects of conservative clinical diagnostics by collecting symptoms via ePRO in addition to intensive diagnostics (CA-125 testing, imaging diagnostics) during follow-up, on survival, time to clinical recurrence and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Between diagnosis and the first follow-up visit after the end of their antineoplastic treatment (systemic therapy or surgical treatment) for ovarian cancer.
* German, English, French, or Italian speaking
* Personal smartphone (iOS or Android system); one of the latest three main versions

Exclusion Criteria:

• Patients whose compliance must be questioned, e.g. due to a psychiatric disorder, private life situation or insufficient knowledge on smartphone use and do not have a suitable caregiver to assist them with symptom reporting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women ≥ 18 years old with a primary ovarian cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Overall survival three years after end of therapy | 3 years
  Overall survival three years after the end of primary therapy / start of follow-up

SECONDARY OUTCOMES:
Time to Recurrence | 3 years
  Time to Recurrence
Total number of tumor relapses | 3 years
  Total number of tumor relapses occurring in the follow-up period
Well-being | 3 years
  Well-being according to the ECOG Performance Status
  GRADE ECOG PERFORMANCE STATUS 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
Amount and frequency of patient data entries | 3 years
  Amount and frequency of patient data entries
Platinum-sensitivity and the patients' platinum free interval (PFI) | 3 years
  Platinum-sensitivity and the patients' platinum free interval (PFI)
Number and type of unplanned hospitalizations and emergencies. | 3 years
  Unplanned hospitalizations and emergencies are defined as additional consultations outside of planned therapy or control visits at the treatment center or with the investigator, as well as unplanned visits to other physicians (e.g., GP) or emergency services.
Symptoms that led to further diagnostic measures and possibly the detection of tumor relapse | 3 years
  Symptoms that led to further diagnostic measures (imaging diagnostics and CA-125 testing) and possibly the detection of tumor relapse

CONTACTS AND LOCATIONS:
Overall Officials: Pius Wyss, Prof.Dr.med, Principal Investigator — Swiss Tumor Institue
Locations (4):
- Switzerland (4):
  - Spital Limmattal Frauenklinik, Schlieren, Canton of Zurich
  - Gynäkologische Onkologie Spital Zollikerberg, Zollikerberg, Canton of Zurich
  - Praxis für Gynäkologie und Geburtshilfe, Zurich
  - Interdisziplinäre Medizin Zürich (IMZ), Zurich